CLINICAL TRIAL: NCT03560245
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study Assessing the Safety, Tolerability and Efficacy of Bryostatin in the Treatment of Moderately Severe to Severe Alzheimer's Disease Subjects Not Receiving Memantine Treatment
Brief Title: A Study of Bryostatin in Moderately Severe to Severe Alzheimer's Disease Subjects Not On Memantine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotrope Bioscience, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTRP101-203
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Bryostatins

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be stratified based on Mini Mental State Exam (MMSE-2) scores 4-9 vs. 10-15 and will be randomized 1:1 to one of two treatment arms: 20µg bryostatin or placebo for twelve weeks (7 doses).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bryostatin 20µg (Experimental): 20µg Bryostatin administered IV over 45 minutes every other week after 2 initial loading doses of 24 micrograms administered weekly. A total of 7 doses administered over 12 weeks.
  Interventions: Drug: Bryostatin
- Placebo (Placebo Comparator): Placebo administered IV over 45 minutes every other weekafter 2 initial doses administered weekly. A total of 7 doses administered over 12 weeks.
  The placebo is a sterile, pyrogen-free, lyophilized powder identical in appearance to the active drug, intended for IV infusion upon reconstitution and dilution.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bryostatin — The investigational drug product, bryostatin, is a sterile, pyrogen-free, lyophilized powder intended for IV infusion upon reconstitution and dilution.
  Arms: Bryostatin 20µg
Other: Placebo — The placebo is a sterile, pyrogen-free, lyophilized powder identical in appearance to the experimental drug
  Arms: Placebo

SUMMARY:
This is a randomized double-blind Placebo-controlled, Phase 2 study comparing bryostatin to placebo for the treatment of moderately severe to severe Alzheimer's disease in subjects not receiving memantine treatment. The study is 15 weeks in duration, including a safety and efficacy evaluation 30 days after the last dose of study drug. Subjects will receive 7 doses of study drug during the study. The primary efficacy endpoint is defined as the change from baseline to Week 13 in the Severe Impairment Battery (SIB) total score.

DETAILED DESCRIPTION:
Eligible subjects will be stratified based on Mini Mental State Exam (MMSE-2) scores 4-9 vs. 10-15 and will be randomized 1:1 to one of two treatment arms: 20µg bryostatin or placebo for twelve weeks. The first two doses of study drug will be a loading dose 20% higher (i.e., 24µg) than the assigned dose and will be administered one week apart. Thereafter, the assigned dose of 20µg will commence with the third dose and be administered every other week. Drug is administered IV by continuous infusion over 45(±5) minutes. Subjects are scheduled to receive seven doses over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from caregiver and subject (if possible) or legally acceptable representative if different from caregiver
2. Male and female subjects 55-85 years of age inclusive
3. Cognitive deficit present for at least 2 years that meet the diagnostic criteria for probable Alzheimer's dementia. The diagnosis must be confirmed at the time of the screening visit
4. MMSE-2 score of 4-15 inclusive (applies to Screening Visit only)
5. Patients must be able to perform at least one item on the SIB and may not have a SIB score >93 at screening
6. Neuroimaging computerized tomography (CT) or Magnetic Resonance Imaging (MRI) within the last 24 months consistent with a diagnosis of probable AD without any other clinically significant co-morbid pathologies. If there has been a significant change in the subject's clinical status since the last imaging study that is not consistent with progression of the subject's AD, an imaging study should be performed to confirm eligibility
7. Reliable caregiver(s) or informant(s) who attends the subject at least an average of 3 hours or more per day for 3 or more days per week and who will agree to accompany the subject to the clinic visits and reliably complete the caregiver questions
8. Adequate vision and motor function to comply with testing
9. If taking an approved cholinesterase inhibitor for treatment of Alzheimer's disease, must be on a stable dose for at least 3 months prior to entry into study and the dose must not change during the study unless a change is required due to an adverse effect of the prescribed medication or a clinically significant change in the patient's status
10. Subjects who are memantine naïve or have been off memantine for at least 30 days prior to initial treatment with study drug
11. Subjects on neuroleptic medications must be on a stable dose for ≥4 weeks (dose adjustments will be permitted)
12. Females participating in the study must meet one the following criteria:

    1. Surgically sterilized (e.g., hysterectomy, bilateral oophorectomy or tubal ligation) for at least 6 months or postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 year) or
    2. If not postmenopausal, agree to use a double method of contraception, one of which is a barrier method (e.g., intrauterine device plus condom, spermicidal gel plus condom) 30 days prior to dosing until 30 days after last dose and have negative human chorionic gonadotropin (β-hCG) test for pregnancy at screening
13. Males who have not had a vasectomy must use appropriate contraception methods (barrier or abstinence) from 30 days prior to dosing until 30 days after last dose
14. In the opinion of the PI subjects should be in reasonably good health over the last 6 months and any chronic disease should be stable -

Exclusion Criteria:

1. Dementia due to any condition other than AD, including vascular dementia (Rosen-Modified Hachinski Ischemic score ≥ 5)
2. Evidence of significant central nervous system (CNS) vascular disease on previous neuroimaging including but not limited to: cortical stroke, multiple infarcts, localized single infarcts in the thalamus, angular gyrus, multiple lacunar infarcts or extensive white matter injury
3. Clinically significant neurologic disease or condition other than AD, such as cerebral tumor, chronic subdural fluid collections, Huntington's Disease, Parkinson's Disease, normal pressure hydrocephalus, or any other diagnosis that could interfere with assessment of safety and efficacy
4. Evidence of clinically significant unstable cardiovascular, pulmonary, renal, hepatic, gastrointestinal, neurologic, or metabolic disease within the 6 months prior to enrollment. . If there is a history of cancer the subject should be clear of cancer for at least 2 years prior to screening. More recent history of basal cell or squamous cell carcinoma and melanoma in situ (Stage 0) may be acceptable after review by the Medical Monitor.
5. Creatinine clearance (CL) of <45ml/min
6. Poorly controlled diabetes, at the discretion of the Principal Investigator
7. Concomitant treatment with NMDA receptor antagonists such as but not limited to memantine or drug combinations containing memantine, dextromethorphan (a cough suppressant), ketamine, phencyclidine (PCP), methoxetamine (MXE), nitrous oxide (N2O) and the following synthetic opioids: penthidine, levorphanol, methadone, dextropropoxyphene, tramadol, and ketobemidone.
8. Use of vitamin E > 400 International Units (IU) per day within 14 days prior to screening
9. Use of valproic acid within 14 days prior to screening
10. Use of an active Alzheimer's vaccine within 2 years prior to screening
11. Use of a monoclonal antibody for treatment of AD within 1 year prior to screening
12. Any medical or psychiatric condition that is likely to require initiation of additional medication or surgical intervention during the course of the study
13. Any screening laboratory values outside the reference ranges that are deemed clinically significant by the PI
14. Use of an investigational drug within 30 days prior to screening
15. Suicidality defined as active suicidal thoughts during the 6 months prior to screening or at Baseline [Type 4 or 5 on C-SSRS], or history of suicide attempt in previous 2 years, or at serious suicide risk in PI's judgment
16. Major psychiatric illness such as current major depression according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition , current or past diagnosis of bipolar disorder, schizophrenia, or any other psychiatric disorder that might interfere with the assessments of safety or efficacy at the discretion of the PI
17. Diagnosis of alcohol or drug abuse within the last 2 years
18. Abnormal laboratory tests that suggest an alternate etiology for dementia. If the patient has prior history of serum B12 abnormality, anemia with hemoglobin ≤10g /dl, thyroid function abnormality, electrolyte abnormality, or positive syphilis serology the patient should be revaluated to determine if these potential causes of dementia have been addressed. Only if these causes have been ruled out as the cause of the dementia can the patient be enrolled.
19. History of prolonged QT or prolonged QT on screening ECG (QTcB or QTcF >499 per central reader)
20. Acute or poorly controlled medical illness: blood pressure > 180 mmHg systolic or 100 mmHg diastolic; myocardial infarction within 6 months; uncompensated congestive heart failure [New York Heart Association (NYHA) Class III or IV]
21. Known to be seropositive for human immunodeficiency virus (HIV)
22. Known to be seropositive for Hepatitis B or C, unless successful curative treatment for Hepatitis C (e.g., Harvoni) has been received and there is documentation that there is no Hep B/C virus detected 3 months after completion of treatment
23. AST or ALT >3x upper limit of normal (ULN) and total bilirubin >2x ULN or International Normalized Ratio (INR) >1.5
24. Prior exposure to bryostatin, or known sensitivity to bryostatin or any ingredient in the study drug
25. Any other concurrent medical condition, which in the opinion of the PI makes the subject unsuitable for the clinical study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tuchman, MD, Study Director — Neurotropebioscience, Inc
Locations (28):
- United States (28):
  - Neuro Pain Medical Center, Fresno, California
  - Nader Pharmacology Research Institute, Los Alamitos, California
  - Syrentis Clinical Research, Santa Ana, California
  - Southern California Research, LLC, Simi Valley, California
  - JEM Research, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Miami Jewish Health / Stein Gerontological Institute, Miami, Florida
  - Phoenix Medical Research, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Bioclinica Research, Orlando, Florida
  - Anchor Neuroscience, Pensacola, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Bioclinica Research, The Villages, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Medical Research & Health Education Foundation, Columbus, Georgia
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Alzheimer's Disease Center, Quincy, Massachusetts
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - Burke Rehabilitation Hospital, White Plains, New York
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Insight Clinical Trials, LLC, Shaker Heights, Ohio
  - Memory Health Center at Summit Research Network, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 111 subjects were randomized, but 3 subjects withdrew prior to receiving treatment. 108 subjects received treatment.
Groups:
- Placebo: Placebo administered IV over 45 minutes every other weekafter 2 initial doses administered weekly. A total of 7 doses administered over 12 weeks.
  The placebo is a sterile, pyrogen-free, lyophilized powder identical in appearance to the active drug, intended for IV infusion upon reconstitution and dilution.
  Placebo: The placebo is a sterile, pyrogen-free, lyophilized powder identical in appearance to the experimental drug
Period: Overall Study
Arm/Group | Bryostatin 20µg | Placebo
Started | 53 | 55
Completed | 48 | 48
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: There were 108 subjects who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bryostatin 20µg | Placebo | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 40 | 45 | 85
Sex: Female, Male [Count of Participants; unit: Participants] — There were 111 randomized subjects, however 3 subjects never received study drug. Population: The Safety Analysis Set (SAS) was defined as all randomized subjects who received any study medication (either partial or completed infusions of bryostatin or placebo).
  Participants
    Female | 29 | 32 | 61
    Male | 24 | 23 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 44 | 47 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 42 | 49 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 55 | 108
Safety Analysis Set [Count of Participants; unit: Participants] — Safety Analysis Set = subjects who received any dose of study drug (either partial or completed infusions of bryostatin or placebo).
  Participants | 53 | 55 | 108

OUTCOME MEASURES:

1. Primary Outcome: Safety: Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Incidence of adverse events (AEs), serious adverse events (SAEs), Adverse event of special interest - myalgia
Time Frame: Baseline through 30 days post end of treatment (up to Day 107)
Population: All participant who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Bryostatin 20µg | Placebo
Number analyzed (Participants) | 53 | 55
Participants | 21 | 10

2. Primary Outcome: Efficacy: The Primary Efficacy Endpoint is Defined as the Change From Baseline to Week 13 in the Severe Impairment Battery (SIB) Total Score in the Full Analysis Set
Description: The Severe Impairment Battery (SIB) assesses cognition in subjects with moderate and severe Alzheimer's disease(AD). Test questions measure attention, language, orientation, memory, praxis, visuospatial ability, construction, social skills, orienting head to name. Non-verbal responses are allowed, thus decreasing the need for language output. Forty questions are included with a total point score range of 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: The change in the SIB Total Score from baseline to Week 13 (Day 91)
Population: The Full Analysis Set (FAS) used for efficacy analyses was defined as all randomized subjects who received at least one dose of study medication and who have at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bryostatin 20µg: Subjects were scheduled to receive seven doses over 12 weeks. The first two doses of study drug were to be a loading dose 20% higher (i.e., 24µg) than the assigned dose and were to be administered one week apart. Thereafter, the assigned dose of 20µg was to commence with the third dose and be administered every other week. The study drug was administered intravenously (IV) by continuous infusion over 45(±5) minutes.
- Placebo: Subjects were scheduled to receive seven doses over 12 weeks. The study drug was administered intravenously (IV) by continuous infusion over 45(±5) minutes.
Arm/Group | Bryostatin 20µg | Placebo
Number analyzed (Participants) | 52 | 54
score on a scale | 1.3 (8.42) | 2.1 (9.22)
Statistical Analysis 1: Comparison: Bryostatin 20µg vs Placebo; Test type: Equivalence — The change from baseline to Week 13 in the SIB total score was summarized descriptively and compared using Analysis of Covariance (ANCOVA) adjusted for baseline SIB total score. If the normality assumption was not met, a non-parametric method or a rank-ANCOVA analysis (i.e., an ANCOVA analysis on rank-transformed data) was to be used; p = 0.3730, t-test, 2 sided

3. Secondary Outcome: The Changes From Baseline at Weeks 5, 9 and 15 in the Severe Impairment Battery (SIB) Total Score in the Full Analysis Set.
Description: The Severe Impairment Battery (SIB) assesses cognition in subjects with Alzheimer's disease. SIB scores at Weeks 5, 9 and the Week 15 follow-up visit will be assessed. Test questions measure attention, language, orientation, memory, praxis, visuospatial ability, construction, social skills, orienting head to name. Non-verbal responses are allowed, thus decreasing the need for language output. Forty questions are included with a total point score range of 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: Weeks 5, 9 and 15 (up to Day 107)
Population: At each timepoint, the number of participants whose data was obtained could vary from the number of subjects enrolled. There were occasions when subjects missed a visit or dropped out of the study, resulting in fewer data captured at that timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bryostatin 20µg | Placebo
Number analyzed (Participants) | 52 | 54
score on a scale
  Week 5: number analyzed (Participants) | 52 | 51
  Week 5 | -0.1 (7.94) | 0.7 (11.0)
  Week 9: number analyzed (Participants) | 49 | 51
  Week 9 | 2.7 (7.18) | 1.4 (8.23)
  Week 15 or early termination: number analyzed (Participants) | 48 | 51
  Week 15 or early termination | 1.6 (9.07) | 2.1 (9.66)

4. Secondary Outcome: The Changes From Baseline at Weeks 5, 9, 13 and 15 in the Severe Impairment Battery (SIB) Total Score for Subjects in the Mini Mental State Exam Version 2 (MMSE-2) 4-9 Stratification Group
Description: The SIB is used to assess cognition in subjects with moderate and severe AD and is a useful outcome measure in advanced stages of disease. It is divided into nine subscales that include attention, language, orientation, memory, praxis, visuospatial ability, construction, social skills, orienting head to name. Non-verbal responses are allowed, thus decreasing the need for language output. Forty questions are included with a point score range of 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: Weeks 5, 9, 13 and 15 (up to Day 107)
Population: The MMSE-2 4-9 stratification group represents Severe Alzheimer's disease. The analysis population at each time point varies because of missed visits and dropouts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bryostatin 20µg | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale
  Week 5: number analyzed (Participants) | 18 | 17
  Week 5 | -3.1 (9.55) | 1.4 (11.1)
  Week 9: number analyzed (Participants) | 16 | 16
  Week 9 | 1.1 (8.98) | 1.1 (13.3)
  Week 13: number analyzed (Participants) | 17 | 15
  Week 13 | -3.6 (7.42) | 1.9 (15.3)
  Week 15/ Early Termination: number analyzed (Participants) | 16 | 15
  Week 15/ Early Termination | -2.6 (9.81) | 0.3 (16.5)

5. Secondary Outcome: The Changes From Baseline at Weeks 5, 9, 13 and 15 in the Severe Impairment Battery (SIB) Total Score for Subjects in the Mini Mental State Exam Version 2 (MMSE-2) 10-15 Stratification Group
Description: Mini Mental State Exam version 2 (MMSE-2) scores between 10 and 15 are representative of moderately severe Alzheimer's disease. The SIB is used to assess cognition in subjects with moderate and severe AD and is a useful outcome measure in advanced stages of disease. It is divided into nine subscales that include attention, language, orientation, memory, praxis, visuospatial ability, construction, social skills, orienting head to name. Non-verbal responses are allowed, thus decreasing the need for language output. Forty questions are included with a point score range of 0-100. Lower scores indicate greater cognitive impairment.
Time Frame: Weeks 5, 9, 13 and 15 (up tp Day 107)
Population: Mini Mental State Exam version 2 (MMSE-2) scores between 10 and 15 are representative of moderately severe Alzheimer's disease. The number of participants at each time point varies because of missed visits and dropouts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bryostatin 20µg | Placebo
Number analyzed (Participants) | 34 | 36
score on a scale
  Week 5: number analyzed (Participants) | 34 | 34
  Week 5 | 1.4 (6.57) | 0.3 (11.1)
  Week 9: number analyzed (Participants) | 33 | 35
  Week 9 | 3.5 (6.13) | 1.5 (4.61)
  Week 13: number analyzed (Participants) | 32 | 33
  Week 13 | 3.9 (7.80) | 2.2 (4.78)
  Week 15/Early Termination: number analyzed (Participants) | 32 | 36
  Week 15/Early Termination | 3.7 (8.03) | 2.8 (4.74)

6. Secondary Outcome: Individual Patient's Slope Over Time in SIB Total Score Evaluated Via Weeks 0, 5, 9, and 13
Description: Severe Impairment Battery (SIB) trend analyses will be assessed for individual patients. SIB scores were evaluated in subjects at various time points during the study. Individual-specific SIB slopes were estimated for all patients over each person's available SIB outcome measures.
Time Frame: Baseline through Week 13 (Day 91)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Bryostatin 20µg | Placebo
Number analyzed (Participants) | 52 | 54
Participants
  Slope > 0 | 29 | 29
  Slope < 0 | 23 | 23
  Slope = 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were defined as an event with onset on or after the first treatment administration. The time duration was 15 weeks, beginning on the date of the first dose, including a period of 30 days after the last study drug treatment.
Arm/Group | Bryostatin 20µg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/55
Serious Adverse Events (participants affected / at risk) | 5/53 | 6/55
Other Adverse Events (participants affected / at risk) | 16/53 | 4/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bryostatin 20µg (N=53) | Placebo (N=55)
Right Distal Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Well-diferentiated invasive colorectal adenocarcino (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bryostatin 20µg (N=53) | Placebo (N=55)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 1 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 6 (6) | 1 (1)

LIMITATIONS AND CAVEATS:
An imbalance in the baseline Severe Impairment Battery (primary endpoint) was observed between the bryostatin treatment group and the placebo group, with the placebo group having an average SIB score higher than the treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03560245/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03560245/SAP_001.pdf